CLINICAL TRIAL: NCT05993130
Title: Kayseri City (Education and Research) Hospital
Brief Title: Evaluation of Patients With Covid-19 Infection in Terms of Severity of Osteoprosis
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Ayşe Güç, physical medicine and rehabilitation, Kayseri Education and Research Hospital
Other Study IDs: Kayseri City Hospital
Record Dates: First submitted 2023-08-14; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Severity of Osteoprosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The patients were not intervened. This is a retrospective study — The patients were not intervened. This is a retrospective study

SUMMARY:
Osteoporosis is a condition characterized by decreased bone strength and an increased risk of fracture. Age, gender, body mass index, fragility fracture history, corticosteroid use, immobilization, smoking and alcohol use, endocrine pathologies besides inflammatory and infectious pathologies can also be effective in the development of osteoporosis. The aim of the study is to evaluate the effect of Covid-19 infection on the development of osteoporosis.

In this study, bone mineral density (BMD) measurements of patients with Covid-19 infection were examined. For this, dual-energy x-ray absorptiometry (DEXA) measurement was used. A total of 55 patients were included in the study and data such as age, height, weight, comorbidities, drugs used, and treatment methods were recorded. Results showed that the time spent in the intensive care unit was associated with the femoral neck T score in DEXA measurements of patients with Covid-19 infection. The use of drugs such as alendronate, zolendronate, denosumab or teriparatide during the treatment process did not have a statistically significant effect on the lumbar and femur T scores.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over the age of 18 who had dexa measurements twice before and after covid, with at least one year between two dexa measurements, and at least one month after covid infection were included in the study.

Exclusion Criteria:

* Under the age of 18, male patients, patients with a diagnosis other than Covid-19 infection that will affect bone metabolism between the two dexa shooting dates before and after covid, patients who use another drug other than covid treatment that will affect bone metabolism between the two dexa shooting dates before and after covid not included in the study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Physically and anatomically female patients were included. There was no difference in the patients included in our study.
Study Population: Between August 2020 and July 2021, two separate excel files were created for the identification numbers of the patients who had DEXA measurements and the identification numbers of the patients who had covid. Then, common ID numbers were found in both excel files in the computer environment. Among these patients, female patients over the age of 18 who had dexa measurements twice before and after covid, with at least one year between two dexa measurements and at least one month after covid infection were included in the study.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Does the severity of osteoporosis increase in patients with Covid-19 infection? | 2020 August 2021 July

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No